CLINICAL TRIAL: NCT02262104
Title: Effects of an Exercise Program for Nursing Home Patients With Dementia - a Six Months Assessor Blind Randomized Controlled Trial
Brief Title: Effects of an Exercise Program for Nursing Home Patients With Dementia
Acronym: EXDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Centre for Ageing and Health (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Elisabeth Wiken Telenius, Research Fellow, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 2012-1150
Record Dates: First submitted 2013-11-23; First posted 2014-10-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Dementia
Keywords: Exercise; dementia; nursing home
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive exercise (Experimental): Intensive strengthening and balance exercises 1 hour twice a week 12 weeks. Lead by physiotherapists.
  Interventions: Behavioral: Intensive exercise
- Control (Placebo Comparator): Control group activities: Social activities one hour twice a week. Light physical activities, reading, conversation, games. Lead by occupational therapist or nursing staff
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intensive exercise — Arm 1: Intervention group. Intensive strength exercise (12RM) for lower limb and balance exercises twice a week for 1 hour. Groups of max 3 participants lead by physiotherapist
  Arms: Intensive exercise
Behavioral: Control — Arm 2: control. Social activity group with light exercise, reading, and games. Lead by occupational therapist or nursing staff
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the effect of an exercise program on nursing home patients with dementia.

DETAILED DESCRIPTION:
The intervention group will be exercising one hour twice a week for 12 weeks. The participants will be doing intensive strength exercises and challenging balance exercises in groups of 4-6. Two physical therapists will be leading the intervention group. The control group will be meeting at the same frequency. Groups of 4-6 will be lead by an occupational therapist. The participants will be doing relaxation exercises, listen to music and social activities such as board games or indoor bowling.

The investigators will carry out three test periods:

* Baseline testing before intervention start
* Post test after 12 weeks of intervention
* Follow-up 12 weeks after post test.

The testing will comprise:

* Physical tests carried out by physiotherapists
* Questionnaires concerning mental health and ADL (activities of daily living)
* Cognition tests
* Cortisol in saliva

ELIGIBILITY:
Inclusion Criteria:

* >55 years old
* Living in nursing home
* Able to stand with help from max 1
* Able to walk 6 meters with or without walking aid

Exclusion Criteria:

* Medically unstable
* Longterm psychotic
* Severe communication problems

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, Principal Investigator — Oslo and Akershus University college of Applied science
Locations (1):
- Oslo and Akershus University College of Applied Sciences, Oslo, Norway

REFERENCES:
- [Derived] Kvael LAH, Bergland A, Telenius EW. Associations between physical function and depression in nursing home residents with mild and moderate dementia: a cross-sectional study. BMJ Open. 2017 Jul 20;7(7):e016875. doi: 10.1136/bmjopen-2017-016875. PMID 28729326
- [Derived] Telenius EW, Engedal K, Bergland A. Long-term effects of a 12 weeks high-intensity functional exercise program on physical function and mental health in nursing home residents with dementia: a single blinded randomized controlled trial. BMC Geriatr. 2015 Dec 3;15:158. doi: 10.1186/s12877-015-0151-8. PMID 26630910
- [Derived] Telenius EW, Engedal K, Bergland A. Effect of a high-intensity exercise program on physical function and mental health in nursing home residents with dementia: an assessor blinded randomized controlled trial. PLoS One. 2015 May 14;10(5):e0126102. doi: 10.1371/journal.pone.0126102. eCollection 2015. PMID 25974049